CLINICAL TRIAL: NCT01367249
Title: Efficacy and Safety of Bromfenac Ophthalmic Solution vs. Placebo for the Treatment of Ocular Inflammation and Pain Associated With Cataract Surgery.
Brief Title: Efficacy of Bromfenac Ophthalmic Solution in Patients Undergoing Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S00124
Record Dates: First submitted 2011-06-01; First posted 2011-06-07 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Pain; Inflammation; Cataract
Keywords: cataract surgery
MeSH Terms: conditions — Pain; Inflammation; Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromfenac Ophthalmic Solution (Experimental): Bromfenac ophthalmic solution 0.07% one drop into study eye, once daily (QD) starting the day before cataract surgery and continued for 14 days post surgery for a total of 16 days.
  Interventions: Drug: Bromfenac Ophthalmic Solution
- Placebo (Placebo Comparator): One drop of placebo into study eye, once daily (QD) starting the day before cataract surgery and continued for 14 days post surgery for a total of 16 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bromfenac Ophthalmic Solution — Sterile ophthalmic solution
  Arms: Bromfenac Ophthalmic Solution
Drug: Placebo — Sterile ophthalmic solution
  Arms: Placebo

SUMMARY:
This is an efficacy study of Bromfenac Ophthalmic Solution in cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age who are scheduled for unilateral cataract surgery

Exclusion Criteria:

* Have known hypersensitivity to bromfenac or to any component of the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multi-center, randomized, double-masked, parallel-group, placebo-controlled study, the first subject was enrolled 05/05/2011 and the last subject exited the study 07/29/2011.
Pre-assignment Details: 440 subjects were enrolled from 39 clinical sites in the United States, of which 416 subjects received at least 1 dose of bromfenac or placebo.
Groups:
- Placebo: One drop of placebo into study eye, once daily (QD) starting the day before cataract surgery and continued for 14 days post surgery for a total of 16 days.
  Placebo: Sterile ophthalmic solution, vehicle of bromfenac ophthalmic solution
Period: Overall Study
Arm/Group | Bromfenac Ophthalmic Solution | Placebo
Started | 222 | 218
Completed | 213 | 202
Not Completed | 9 | 16
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Other | 3 | 10

BASELINE CHARACTERISTICS:
Population: Intent to treat population (ITT), all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromfenac Ophthalmic Solution | Placebo | Total
Number analyzed (Participants) | 222 | 218 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.70) | 68.5 (9.68) | 68.5 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 146 | 287
  Male | 81 | 72 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 17 | 39
  White | 167 | 162 | 329
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 31 | 59
Region of Enrollment [Number; unit: participants]
  United States | 222 | 218 | 440
Iris Color (Study Eye) [Number; unit: participants]
  Blue | 57 | 65 | 122
  Brown | 109 | 93 | 202
  Gray | 1 | 5 | 6
  Green | 24 | 21 | 45
  Hazel | 31 | 33 | 64
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Ocular Inflammation
Description: The proportion of subjects who had cleared ocular inflammation summed ocular inflammation score (SOIS) of grade 0 by Day 15.
Time Frame: Day 15
Population: LOCF Analysis, ITT Population
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bromfenac Ophthalmic Solution | Placebo
Number analyzed (Participants) | 222 | 218
Number analyzed (eyes) | 222 | 218
eyes | 108 | 53

2. Secondary Outcome: Ocular Pain
Description: The proportion of subjects who were free of ocular pain at Day 1. Pain Free defined as a score of "None" on the pain scale of the Ocular Comfort Grading Assessment in the subject diary.
Time Frame: Day 1
Population: LOCF Analysis, ITT Population
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bromfenac Ophthalmic Solution | Placebo
Number analyzed (Participants) | 222 | 218
Number analyzed (eyes) | 222 | 218
eyes | 175 | 108

ADVERSE EVENTS:
Time Frame: 16 days
Arm/Group | Bromfenac Ophthalmic Solution | Placebo
Serious Adverse Events (participants affected / at risk) | 3/212 | 4/204
Other Adverse Events (participants affected / at risk) | 29/212 | 54/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromfenac Ophthalmic Solution (N=212) | Placebo (N=204)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) — Subject recovered and the AE resolved
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Eye operation complication (Eye disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Asthenia (Nervous system disorders) | 0 (0) | 1 (1)
Myocarial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromfenac Ophthalmic Solution (N=212) | Placebo (N=204)
Anterior Chamber Inflammation (Eye disorders) | 10 (10) | 18 (18)
Conjunctival Hyperemia (Eye disorders) | 3 (3) | 15 (15)
Eye Pain (Eye disorders) | 12 (12) | 20 (20)
Photophobia (Eye disorders) | 4 (4) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other